CLINICAL TRIAL: NCT01663870
Title: Integrating Technology and Navigation to Improve Survivorship Care in Underserved Populations
Brief Title: Technology and Navigation to Improve Survivorship Care
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-0450
Record Dates: First submitted 2012-08-08; First posted 2012-08-13 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
Keywords: Cancer Prevention; Breast cancer survivors; Cancer survivorship clinic; eHealth technology; Internet; HealthATM website; Questionnaire; Clinic stakeholders; Clinic nurses; Physicians; Case managers; Oncology patient navigators; Audio recorded interviews
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer Survivors: Patients in the LBJ General Hospital Cancer Survivorship Clinic.
  Interventions: Behavioral: Audio Recorded Interviews; Other: Website Session; Behavioral: Questionnaire
- Clinic Stakeholders: Survivorship clinic stakeholders include clinic nurses, physicians, case managers, oncology patient navigators currently working with those in active treatment, information technology support professionals from the Harris County Hospital District (HCHD).
  Interventions: Behavioral: Audio Recorded Interviews; Behavioral: Focus Group Session; Other: Website Session

INTERVENTIONS:
Behavioral: Audio Recorded Interviews — Audio recorded interview at beginning of visit and after using HealthATM website.
Behavioral: Focus Group Session — Focus group session taking 60-90 minutes.
  Groups: Clinic Stakeholders
Other: Website Session — 10-15 minute session with the HealthATM website.
Behavioral: Questionnaire — Questionnaire completion at end of audio recorded interview taking about 5 minutes.
  Other Names: Survey
  Groups: Breast Cancer Survivors

SUMMARY:
The goal of this research study to learn about breast cancer survivorship and possible ways to improve breast cancer survivorship programs using technology.

Objectives:

Objective 1: Assess breast cancer survivors on the acceptability of and preferences for the integration of patient navigation and an eHealth technology platform to improve care in the Survivorship Clinic at Lyndon B. Johnson Hospital.

Objective 2: Assess clinic stakeholders acceptability of and preferences for the integration of patient navigation and an eHealth technology platform to improve care for breast cancer patients in the Survivorship Clinic at Lyndon B. Johnson Hospital.

DETAILED DESCRIPTION:
Breast Cancer Survivors:

If patient agrees to take part in this study, they will visit the cancer survivorship clinic where the following tests and procedures will be performed:

* Patient will have a 30-60 minute interview where they will be asked about cancer-related informational needs, feelings about survivorship care plans, and preferred methods of communication with survivorship clinic staff.
* Patient will be asked about whether they would use the internet and other technologies (such as text messages for appointment reminders) as tools in breast cancer survivorship.
* Patient will use a web-based tool called HealthATM. HealthATM is a website that is designed to provide information and tools to help patients better manage their health. After 10-15 minute session with the website, patient will be asked about how easy the website was to use and other questions about their session.
* Patient will complete a short questionnaire at the end of the interview asking about personal characteristics, how involved they are in their health care, and their attitudes towards the HealthATM website. It should take about 5 minutes to complete this questionnaire.

All interviews will be audiorecorded. All audio recordings will be kept for 5 years and then destroyed. All interview data will be stored in password-protected computers and/or locked file cabinets. There will be no personal identifying information connected to patient's interview answers.

Length of Study:

All of the study procedures will take place at one visit. The visit should last about 60 minutes.

This is an investigational study.

Up to 40 participants will be enrolled in this study. All will be enrolled at LBJ General Hospital.

Clinic Stakeholders:

If clinic staff agree to take part in this study, the following tests and procedures will be performed:

* Clinic staff will take part in a 60-90 minute focus group session where they will be asked about their feelings about survivorship care plans and if they think web-based eHealth programs would be helpful as tools in breast cancer survivorship.
* Clinic staff will be asked about any challenges and barriers they feel are facing the survivorship programs at LBJ.
* Clinic staff will use a web-based tool called HealthATM. HealthATM is a website that provides information and tools to help patients better manage their health. After a 10-15 minute session with the website, they will be asked about how easy the website was to use and other questions about their session.

All focus group sessions will be audiorecorded. All audio recordings will be kept for 5 years and then destroyed. All focus group data will be stored in password-protected computers and/or locked file cabinets. There will be no personal identifying information connected to your focus group answers.

Length of Study:

All of the study procedures will take place at one visit. The visit should last about 60 minutes.

This is an investigational study.

Up to 40 stakeholders will be enrolled in this study. All will be enrolled at LBJ General Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-years or older (survivors and stakeholders)
2. Ability to read and speak English or Spanish (survivors)
3. Ability to read and speak English (stakeholders)
4. Active patient at the LBJ General Hospital Survivorship Clinic (survivors only)
5. Previous cancer diagnosis with no evidence of recurrence at 3 years or greater following initial diagnosis (survivors only)
6. Harris County Hospital District employee offering clinical or administrative support to the LBJGH Cancer Survivorship Clinic (stakeholders only)
7. Cancer survivors who are at least 6 months from diagnosis

Exclusion Criteria:

1) None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer survivors and stakeholders at LBJ General Hospital Cancer Survivorship Clinic in Houston, Texas
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-02; Primary Completion 2020-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Interview Study of Breast Cancer Survivorship Programs Using Technology | 1 day
  Breast cancer survivors and clinic staff surveys analyzed regarding acceptability of, and preferences for integration of patient navigation and an eHealth technology platform. Focus group and interview transcripts analyzed using ATLAS.ti qualitative analysis software. To analyze these data, constant comparative method used to conduct thematic analysis of transcribed data. As secondary check of breast cancer survivor data, calculation of descriptive statistics for measures administered to survivors following interview (frequencies, means, and standard deviations) including Patient Activation Measure and Systems Usability Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Peterson, MPH, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Lyndon B. Johnson Hospital, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org